CLINICAL TRIAL: NCT03736304
Title: The Effect of Automated Electronic Alert for Acute Kidney Injury on the Outcomes of Hospitalized Patients: a Single Center Randomized Controlled Trial.
Brief Title: The Effect of Automated Electronic Alert for Acute Kidney Injury on the Outcomes of Hospitalized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2018-SR-180
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Acute Kidney Injury; Outcomes; Early Diagnosis
MeSH Terms: conditions — Acute Kidney Injury; Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: All study investigators and participants were blinded to patients randomization status.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Placebo Comparator): Patients will receive standard clinical care by the doctor in charge.
  Interventions: Other: Usual care
- AKI alert (Experimental): An AKI alert will send to the the doctor in charge. The team of nephrologists would give suggestions if the doctor in charge need a renal consultation.
  Interventions: Device: AKI alert

INTERVENTIONS:
Device: AKI alert — An AKI alert will send to the doctor in charge. The team of nephrologists would give suggestions if the doctor in charge need a renal consultation.
  Arms: AKI alert
Other: Usual care — Patients will receive standard clinical care by the doctor in charge.
  Arms: Usual care

SUMMARY:
Acute kidney injury (AKI) is a common disease, but diagnosis is usually delayed or missed in hospitalized patients. The automated electronic alert for AKI may help to improve the outcomes of these patients through identifying all cases of AKI early. Therefore, the investigators conduct a randomly controlled study to test whether automated electronic alert for AKI could improve the outcomes of hospitalized patients.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common disease, but diagnosis is usually delayed or missed in hospitalized patients. The automated electronic alert for AKI may help to improve the outcomes of these patients through identifying all cases of AKI early. Therefore, the investigators conduct a randomly controlled study to test whether automated electronic alert for AKI could improve the outcomes of hospitalized patients.

The patients were randomly divided into two groups:

Usual care : patients will receive standard clinical care by the primary physicians AKI alert : an AKI alert will be sent to the doctor in charge. The team of kidney experts would give a suggestion if the doctor in charge need a renal consultation.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adult patients with an Alert for AKI(based on KDIGO guidelines)

Exclusion Criteria:

* Patients already having eGFR<15ml/min/1.73m2 or receiving renal replacement therapy for AKI at the time of alert.
* Patients already having a AKI before admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4536 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Estimated glomerular filtration rate changed within 7 days | within 7 days diagnosed with AKI
  Medical record

SECONDARY OUTCOMES:
seven-day mortality | within 7 days diagnosed with AKI
  Medical record
30-day mortality | within 30 days diagnosed with AKI
  Medical record
1-year mortality | within 1 year diagnosed with AKI
  telephone follow-up
receiving renal replacement therapy at seventh day | 7 days
  Medical record
receiving renal replacement therapy at 30th day | 30 days
  telephone follow-up
receiving renal replacement therapy at 1 year | 1 year
  telephone follow-up
the rate of stage 2 AKI | within 7 days diagnosed with AKI
  Medical record
the rate of stage 3 AKI | within 7 days diagnosed with AKI
  Medical record
the rate of AKI recovery at 90 day | 90 days
  telephone follow-up
the rate of timely-recognition of AKI | 3 days
  Medical record
the interventions for AKI | within 7 days diagnosed with AKI
  Medical record
Follow-up rate after discharge | 1 year
  telephone follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Huijuan Mao, PhD,MD, Principal Investigator — Department of Nephrology, The First Affiliated Hospital of Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Wu B, Li L, Cheng X, Yan W, Liu Y, Xing C, Mao H. Propensity-score-matched evaluation of under-recognition of acute kidney injury and short-term outcomes. Sci Rep. 2018 Oct 11;8(1):15171. doi: 10.1038/s41598-018-33103-9. PMID 30310097
- [Background] Yang L, Xing G, Wang L, Wu Y, Li S, Xu G, He Q, Chen J, Chen M, Liu X, Zhu Z, Yang L, Lian X, Ding F, Li Y, Wang H, Wang J, Wang R, Mei C, Xu J, Li R, Cao J, Zhang L, Wang Y, Xu J, Bao B, Liu B, Chen H, Li S, Zha Y, Luo Q, Chen D, Shen Y, Liao Y, Zhang Z, Wang X, Zhang K, Liu L, Mao P, Guo C, Li J, Wang Z, Bai S, Shi S, Wang Y, Wang J, Liu Z, Wang F, Huang D, Wang S, Ge S, Shen Q, Zhang P, Wu L, Pan M, Zou X, Zhu P, Zhao J, Zhou M, Yang L, Hu W, Wang J, Liu B, Zhang T, Han J, Wen T, Zhao M, Wang H; ISN AKF 0by25 China Consortiums. Acute kidney injury in China: a cross-sectional survey. Lancet. 2015 Oct 10;386(10002):1465-71. doi: 10.1016/S0140-6736(15)00344-X. PMID 26466051
- [Background] Wilson FP, Shashaty M, Testani J, Aqeel I, Borovskiy Y, Ellenberg SS, Feldman HI, Fernandez H, Gitelman Y, Lin J, Negoianu D, Parikh CR, Reese PP, Urbani R, Fuchs B. Automated, electronic alerts for acute kidney injury: a single-blind, parallel-group, randomised controlled trial. Lancet. 2015 May 16;385(9981):1966-74. doi: 10.1016/S0140-6736(15)60266-5. Epub 2015 Feb 26. PMID 25726515
- [Derived] Li T, Wu B, Li L, Bian A, Ni J, Liu K, Qin Z, Peng Y, Shen Y, Lv M, Lu X, Xing C, Mao H. Automated Electronic Alert for the Care and Outcomes of Adults With Acute Kidney Injury: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2351710. doi: 10.1001/jamanetworkopen.2023.51710. PMID 38241047